CLINICAL TRIAL: NCT00527930
Title: Phase II Trial of Oxaliplatin in Combination With S-1(SOX) in Patients With Recurrent or Metastatic Breast Cancer (MBC) Previously Treated With or Resistant to an Anthracycline and Taxane
Brief Title: Phase II Trial of Oxaliplatin in Combination With S-1(SOX) in Patients With Recurrent or Metastatic Breast Cancer
Acronym: TORCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Cancer Study Group (Other); National Cancer Center, Korea (Other Government); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-BR-0703, H-0706-009-209
Record Dates: First submitted 2007-09-08; First posted 2007-09-11 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Oxaliplatin; S1
MeSH Terms: conditions — Breast Neoplasms | interventions — titanium silicide; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TS-1 and Eloxatin — S-1 80 mg/m2/day on day 1-14 Oxaliplatin 130 mg/m2 IV for 2 hour on day 1 Every 3 week
  Number of Cycles: until progression or unacceptable toxicity

SUMMARY:
Phase II trial of oxaliplatin in combination with S-1(SOX) in patients with recurrent or metastatic breast cancer (MBC) previously treated with or resistant to an anthracycline and taxane

DETAILED DESCRIPTION:
The main purpose of this study is to find out the efficacy and safety profile of TS-1 with oxaliplatin in previously anthracycline and taxane pretreated patients.

ELIGIBILITY:
Inclusion Criteria:

* M/F age ≥ 18
* Metastatic(TxNxM1) or inoperable locally recurrent breast cancer(rT4NxM0) after taxane & anthracycline therapy
* Measurable disease (RECIST) : A patient with at least one measurable lesion of which the diameter is confirmed to be 10mm in spiral CT or multidetector CT (MD CT), or 20 mm or longer in conventional CT
* No prior treatment with S-1, capecitabine, platinum In metastatic setting
* Must have received an anthracycline and taxane in adj. or metastatic settings (concurrent, sequential, or combined with other drugs)
* For taxanes (Paclitaxel (P) / Docetaxel (D))

  1. Must have progressed while or after receiving P or D (Patients who relapse within 12 months of completing adjuvant chemotherapy containing an anthracycline and a taxane, do not require prior chemotherapy for metastatic disease)
  2. Only 1 adjuvant regimen permitted (neoadjuvant immediately followed by surgery and immediately followed by adj. is permitted)
* For anthracyclines

  1. Progressed while on anthracycline treatment, with or without initial response or
  2. Have received an adequate course of anthracyclines defined as follows:

  <!-- -->

  1. Adj.: Must have received a standard regimen (doxorubicin ≥ 240 mg/m2 or ≥ 360 mg/m2 epirubicin or equivalent)
  2. Metastatic: Must have received a standard regimen(doxorubicin ≥300mg/m2 or equivalent)
* Not candidate for Herceptin
* ECOG PS ≤ 2
* Completion of all prior chemotherapy ≥ 3 wks prior to enrol
* Completion of hormonal therapy 2 wks prior to enroll
* Resolution of all clinically significant toxic effects (excluding alopecia and sensory neuropathies) of any prior surgery or therapy to grade ≤ 1 (NCI CTCAE 3.0), for peripheral neuropathy grade ≤ 2 (NCI CTCAE 3.0), or to within the limits listed in the specific inclusion/exclusion criteria
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
* Informed consent obtained.

Exclusion Criteria:

* WOCBP(woman of child bearing potential) unwilling to use acceptable method to avoid pregnancy
* Breast feeding or pregnant women
* Patients with Hx of symptomatic brain or leptomeningeal involvement (eligible if asymptomatic 2weeks after proper radiation therapy)
* ≥grade 3 neuropathy currently
* Hx of second malignancy except adequately treated basal or squamous skin ca or CIS of cervix. Adequately treated contralateral breast ca with DF >5 yrs prior to this study is permitted
* MI, unstable angina, CABG, clinically significant arrhythmia within 6 mo
* Hx of inflammatory bowel disease or chronic diarrhea,
* ANC < 1500, Plt < 100K, Hb <9.0
* Ccr < 60 ml/min or creatinine >1.5
* Bil > 1.5 x UNL, AST/ALT ≥ 2.5xUNL if hepatic meta + > 5xUNL)
* History of hypersensitivity to 5-FU, platinum, or to compounds with similar chemical structures
* More than 3 prior chemotherapy for metastatic or recurrent disease or prior treatment with S-1, capecitabine or any platinum analogs in metastatic setting (5-FU combine with other agent in metastatic setting is allowed_ ex) CMF, FAC)
* Her2(+) pts who are candidates for Herceptin
* prior surgery within 4 week
* participate in other clinical trials within 4 week
* prior radiation therapy within 2 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Response Rate | TTP, OS

SECONDARY OUTCOMES:
- To determine the time to progression - To determine the response duration - To determine the overall survival - To determine toxicities - To determine the pharmacogenomic predictor (association study) | PFS, OS

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- See also: Korean Cancer Study Group — http://www.kcsg.org/
- See also: Seoul National University Hospital Clinical Trial Center — http://cris.snuh.org